CLINICAL TRIAL: NCT03384732
Title: Development of a Core Set of the International Classification of Functioning, Disability and Health (ICF) for Geriatric Patients in Primary Care
Brief Title: Development of an ICF Core Set for Geriatric Patients in Primary Care
Acronym: ICF
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, johanna tomandl, Principal Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: 01GY1605
Record Dates: First submitted 2017-12-12; First posted 2017-12-27 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Old and Very Old People; Independent Living; Functioning
Keywords: community-dwelling elderly; ICF; core set development; geriatric; functioning; health; ageing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The sum of medical interventions can do more harm than good. Supporting patients' resources instead of combating disease might effectively help reducing "too much medicine". A first step to approach this goal would be to have a classification tool that captures the essential features of a meaningful human life, namely body functions, activities, and participation. The International Classification of Functioning, Disability and Health (ICF) is the perfect framework to distinguish between necessary and unnecessary medical interventions by offering descriptions of outcomes of medical and non-medical interventions. However, though adequate and comprehensive in theory, it is impracticable in a primary care setting. Therefore, a core set of the ICF for the old and very old in primary care is needed. Four preparatory studies according to the international development guideline will be carried out: a systematic literature review to capture the research perspective, a qualitative study to assess the patients' perspective, an experts' survey and an empirical multicenter study to detect the clinical perspective.

DETAILED DESCRIPTION:
The systematic literature review captures the perspective of researchers on functioning of community dwelling people aged 75 years and older. Different literature databases will be searched combining search terms referring to community dwelling elderly and to functioning. Two investigators will independently screen the abstracts and titles for eligibility. In reviewing the full articles, the underlying concepts that are contained in the measures and in the article text will be identified, and then linked to the ICF categories using established linking rules. A frequency analysis will be conducted on the linked categories. The ICF categories that are identified in at least 5% of all publications will be included in the list of candidate categories.

The qualitative study aims to identify which aspects of functioning, environmental and personal factors are most important to community dwelling people aged 75 years and older. Participants will be provided with a camera for one week to take pictures of activities they are no longer able to perform or activities they still perform well. On the basis of these pictures, individual interviews and focus groups will be conducted. Meaningful concepts will be identified and linked to the ICF categories.

The expert survey aims to gather opinions of experts on aspects of functioning and environmental factors that are relevant for community dwelling people aged 75 years and older. Meaningful concepts will be identified and linked to the ICF categories.

The empirical multicenter study aims to identify the most common problems experienced by community-dwelling people aged 75 and older using clinical assessments. A health professional will conduct semi-structured interviews based on the extended ICF checklist. This is a selection of 125 categories that are considered to be most important for clinical practice. This list is extended by other categories thought to be sensitive to functioning in old age.

ELIGIBILITY:
Systematic review:

Inclusion criteria:

* conducted in the EU, EFTA countries, Australia, New Zealand, USA, Canada
* published in a peer-review journal
* published since 2007
* RCT, controlled clinical trial, cross-sectional study, observational study, qualitative study

Exclusion criteria:

* studies which are solely based on one certain disease
* studies which are solely based on one ethnic group
* studies with hospitalized participants

Qualitative study/empirical multicenter study:

Inclusion criteria:

* community-dwelling people aged 75 years and older

Exclusion criteria:

* people with dementia
* people living in nursing homes
* people in palliative care

Expert survey:

Inclusion criteria

* General practitioners, geriatricians and caregivers with at least two years of professional experience in ambulatory care.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling people aged 75 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Most common health issues of community-dwelling elderly reported in scientific literature (systematic literature review) | 07/2017-10/2018
  The primary outcome will be a core set containing relevant ICF categories from the researchers' perspective.
ADL abilities and disabilities of community-dwelling elderly reported by community-dwelling elderly in semi-structured interviews and focus groups (qualitative study) | 06/2017-01/2018
  The primary outcome will be a core set containing relevant ICF categories from the patients' perspective.
ADL abilities and disabilities of community-dwelling elderly reported by experts in an online survey (expert survey) | 06/2018-04/2019
  The primary outcome will be a core set containing relevant ICF categories from the experts' perspective.
Most common health issues of community-dwelling elderly assessed by the extended ICF checklist (empirical multicenter study) | 04/2018-09/2018
  The primary outcome will be a core set containing relevant ICF categories from the clinical perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kühlein, Prof. Dr., Study Chair — Universitätsklinikum Erlangen, Institute of General Practice
Locations (1):
- Universitätsklinikum Erlangen, Institute of General Practice, Erlangen, Germany

REFERENCES:
- [Background] Selb M, Escorpizo R, Kostanjsek N, Stucki G, Ustun B, Cieza A. A guide on how to develop an International Classification of Functioning, Disability and Health Core Set. Eur J Phys Rehabil Med. 2015 Feb;51(1):105-17. Epub 2014 Apr 1. PMID 24686893
- [Derived] Tomandl J, Heinmuller S, Selb M, Graessel E, Freiberger E, Kuhlein T, Hueber S, Book S, Gotthardt S. Laying the foundation for a Core Set of the International Classification of Functioning, Disability and Health for community-dwelling older adults in primary care: relevant categories of their functioning from the research perspective, a scoping review. BMJ Open. 2021 Feb 17;11(2):e037333. doi: 10.1136/bmjopen-2020-037333. PMID 33597130
- [Derived] Book S, Ulbrecht G, Tomandl J, Kuehlein T, Gotthardt S, Freiberger E, Graessel E. Laying the foundation for an International Classification of Functioning, Disability and Health Core Set for community-dwelling elderly adults in primary care: the clinical perspective identified in a cross-sectional study. BMJ Open. 2020 Nov 23;10(11):e038434. doi: 10.1136/bmjopen-2020-038434. PMID 33234626
- [Derived] Tomandl J, Book S, Gotthardt S, Heinmueller S, Graessel E, Freiberger E, Kuehlein T, Hueber S, Hoyer S. Laying the foundation for a core set of the International Classification of Functioning, Disability and Health for community-dwelling adults aged 75 years and above in general practice: a study protocol. BMJ Open. 2018 Aug 5;8(8):e024274. doi: 10.1136/bmjopen-2018-024274. PMID 30082366